CLINICAL TRIAL: NCT07012876
Title: Effectiveness of a Guided Mental Health Chatbot STARS for Youth Living in Lithuania: a Randomized Controlled Trial
Brief Title: Effectiveness of a Guided Mental Health Chatbot for Youth Living in Lithuania
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vilnius University (Other)
Collaborators: World Health Organization (Other)
Responsible Party: Principal Investigator, Evaldas Kazlauskas, Professor in clinical psychology, Vilnius University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: (1.13E)250000-KT-56/ERC0004137
Record Dates: First submitted 2025-05-16; First posted 2025-06-10 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Symptoms of Depression and Anxiety
Keywords: Intervention; Chatbot; Mental health; Youth; STARS; Effectiveness
MeSH Terms: conditions — Depression; Anxiety Disorders; Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The intervention group will get a guided mental health chatbot STARS.
  Interventions: Behavioral: STARS (Scalable Technology for Adolescents and youth to Reduce Stress)
- Control group (Other): The control group will receive basic psychoeducation. The content of the psychoeducation is very similar to the content of session 2 of the STARS chatbot and includes psychoeducation about emotions, a personal story about a fictional character who talks about her emotions, and information about where to access mental health support. It also includes a list of organizations and clinics providing mental health care in Lithuania.
  Interventions: Behavioral: Basic psychoeducation

INTERVENTIONS:
Behavioral: STARS (Scalable Technology for Adolescents and youth to Reduce Stress) — The intervention is a guided mental health chatbot - STARS - developed by the World Health Organization (WHO). It consists of 10 sessions which include: Introduction (1), Psychoeducation (2), Emotion Regulation (3, 4), Behavior Activation (5, 6), Managing Problems (7), Supportive Self-talk (8, 9), and Relapse Prevention (10). Each session consists of psychoeducation and exercise parts. Trained and supervised non-specialists (called e-helpers) provide weekly calls (five calls lasting approximately 15 minutes) to support participants individually and increase motivation and adherence to the intervention.
  Arms: Intervention group
Behavioral: Basic psychoeducation — The control group will receive basic psychoeducation. The content of the psychoeducation is very similar to the content of session 2 of the STARS chatbot and includes psychoeducation about emotions, a personal story about a fictional character who talks about her emotions, and information about where to access mental health support. It also includes a list of organizations and clinics providing mental health care in Lithuania.
  Arms: Control group

SUMMARY:
The study aims to assess the effectiveness of a guided mental health chatbot called "Scalable Technology for Adolescents and youth to Reduce Stress (STARS)", adapted for youth living in Lithuania.

DETAILED DESCRIPTION:
The intervention is a guided mental health chatbot STARS developed by the World Health Organization (WHO). It consists of 10 sessions which include: Introduction (1), Psychoeducation (2), Emotion Regulation (3, 4), Behavior Activation (5, 6), Managing Problems (7), Supportive Self-talk (8, 9), and Relapse Prevention (10). Each session consists of psychoeducation and exercise parts. Trained and supervised non-specialists (called e-helpers) provide weekly calls (five calls lasting approximately 15 minutes) to support participants individually.

The effect of the intervention will be compared against a control group which receives enhanced usual care.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18-25 years
* Understanding the Lithuanian language
* Having access to a device for intervention delivery
* Experiencing moderate levels of psychological distress (a cut-off score of 8 as measured with Kessler-6)

Exclusion Criteria:

* People at imminent risk of suicide
* People currently experiencing a psychotic episode
* People currently experiencing interpersonal violence
* Current dependency on alcohol/drugs

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 262 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Changes in The Patient Health Questionnaire-9 | Baseline, eight weeks after baseline, three months after baseline
  Changes in symptoms of depression are measured. The Patient Health Questionnaire-9 (PHQ-9, Kroenke et al., 2001) is a self-report measure comprising 9 items about symptoms of depression. All items are answered on a 4-point Likert scale that ranges from 0 (not at all) to 3 (nearly every day). A higher score indicates more pronounced symptoms. In the Lithuanian sample, the PHQ-9 had a good internal consistency with Cronbach's α of 0.85 (Nomeikaite et al., 2023).
Changes in The Generalized Anxiety Disorder-7 | Baseline, eight weeks after baseline, three months after baseline
  Changes in symptoms of anxiety are measured. The Generalized Anxiety Disorder-7 (GAD-7, Spitzer et al., 2006) is a self-report measure comprising 7 items about symptoms of anxiety. All items are answered on a 4-point Likert scale that ranges from 0 (not at all) to 3 (nearly every day). A higher score indicates more pronounced symptoms. In the Lithuanian sample, the GAD-7 had a good internal consistency with Cronbach's α of 0.91 (Nomeikaite et al., 2023).

SECONDARY OUTCOMES:
Changes in Kessler-6 | Baseline, eight weeks after baseline, three months after baseline
  Kessler-6 is used as a screener with a cut-off score of 8, which is commonly used to indicate moderate levels of psychological distress. Also, changes in psychological distress are measured. Kessler-6 (K6, Kessler et al., 2002) is a self-report measure comprising 6 questions about psychological distress. All items are answered on a 5-point Likert scale that ranges from 0 (none of the time) to 4 (all of the time). A higher score indicates more pronounced symptoms. Previous studies have shown good psychometric properties of the Kessler-6 (Cronbach α = 0.86) (Ferro, 2019).
Changes in The Brief Adjustment Disorder Measure-8 | Baseline, eight weeks after baseline, three months after baseline
  Changes in symptoms of adjustment disorder are measured. The Brief Adjustment Disorder Measure-8 (ADNM-8, Kazlauskas et al., 2018) is a self-report measure comprising 8 items about symptoms of adjustment disorder. All items are answered on a 4-point Likert scale that ranges from 1 (never) to 4 (often). A higher score indicates more pronounced symptoms. In the Lithuanian sample, the ADNM-8 had a good internal consistency with Cronbach's α of 0.93 (Kazlauskas et al., 2023).
Changes in The SIDAS | Baseline, eight weeks after baseline, three months after baseline
  Changes in suicidal ideation are measured. The SIDAS (Van Spijker et al., 2014) is a self-report measure comprising 5 questions about suicidal ideation. All items are answered on a 10-point Likert scale that ranges from 0 (never, no control, not close at all, not at all) to 10 (always, full control, made an attempt, extremely). A higher score indicates more pronounced symptoms. In the Lithuanian sample, the SIDAS had a good internal consistency with Cronbach's α of 0.93 (Skruibis et al., 2022).
Changes in The WHODAS 2.0 | Baseline, eight weeks after baseline, three months after baseline
  Changes in functioning are measured. The WHODAS 2.0 (Ustun et al., 2010) is a self-report measure comprising 12 questions about functioning. All items are answered on a 5-point Likert scale that ranges from 0 (none) to 4 (extreme or cannot do). A higher score indicates more pronounced symptoms. Previous studies have shown good psychometric properties of the WHODAS 2.0 (Cronbach α = 0.96) (Saltychev et al., 2021).
Changes in The World Health Organization Well-being Index-5 | Baseline, eight weeks after baseline, three months after baseline
  Changes in psychological well-being are measured. The World Health Organization Well-being Index-5 (WHO-5, Bech, 2004) is a self-report measure comprising 5 items about psychological well-being. All items are answered on a 5-point Likert scale that ranges from 0 (at no time) to 4 (all of the time). A higher score indicates more pronounced psychological well-being. In the Lithuanian sample, the WHO-5 had a good internal consistency with Cronbach's α of 0.87 (Nomeikaite et al., 2023).
Changes in Internalized Stigma of Mental Illness | Baseline, eight weeks after baseline, three months after baseline
  Changes in internalized stigma of psychological difficulties (the term of psychological difficulties instead of mental illness is used in this study) are measured. The Internalized Stigma of Mental Illness-Brief Version (ISMI-10, Boyd et al., 2014) is a self-report measure comprising 10 items about internalized stigma of psychological difficulties. All items are answered on a 4-point Likert scale that ranges from 1 (strongly disagree) to 4 (strongly agree). A higher score indicates more pronounced internalized stigma of psychological difficulties. Previous studies have shown good psychometric properties of the ISMI-10 (Cronbach's α = .75-.81) (Boyd et al., 2014).
Changes in Self-Stigma of Seeking Help | Baseline, eight weeks after baseline, three months after baseline
  Changes in stigma of self-stigma of seeking help are measured. The Self-Stigma of Seeking Help-Ultra-Brief Version (SSOSH-3, Brenner et al., 2021) is a self-report measure comprising 3 items about self-stigma of seeking help. All items are answered on a 5-point Likert scale that ranges from 1 (strongly disagree) to 5 (strongly agree). A higher score indicates more pronounced self-stigma of seeking help. Previous studies have shown good psychometric properties of the SSOSH-3 (Cronbach's α = .82-.87) (Brenner et al., 2021).
Changes in The Client Services Receipt Inventory | Baseline, three months after baseline
  Changes in client service are measured. The Client Services Receipt Inventory (CSRI, Beeacham and Knapp, 2001) is a self-report measure comprising questions about client service. The CSRI covers a broad range of services that may be utilized, including primary and secondary care services, other services, and informal care.
Changes in The EQ-5D-5L | Baseline, eight weeks after baseline, three months after baseline
  Changes in health are measured. The EQ-5D-5L (EuroQol Research Foundation, 2019) is a self-report measure comprising 5 items about health. All items are answered on a 5-point Likert scale that ranges from 1 (I have no problems or similar) to 5 (I am unable or similar). A higher score indicates more pronounced symptoms. Convergent validity was demonstrated by a correlation between EQ-5D-5L and the WHO-5, (r = .43, P < .001) (Janssen et al. 2013).

OTHER OUTCOMES:
International Trauma Exposure Measure before intervention | Baseline
  Number and type of traumatic events before intervention are measured. International Trauma Exposure Measure (ITEM, Hyland et al., 2021) is a self-report measure comprising of 21 items. All items are answered on a dichotomous scale (yes/no). A higher score indicates higher number of traumatic events experienced. ITEM will be used as a predictor in the analysis.
The International Trauma Questionnaire before intervention | Baseline
  Symptoms of post-traumatic stress disorders before intervention are measured. International Trauma Questionnaire (ITQ, Cloitre et al., 2018) is a self-report measure comprising 18 items. All items are answered on a 5-point Likert scale that ranges from 0 (not at all) to 4 (extremely). A higher score indicates more pronounced symptoms. ITQ will be used as a predictor in the analysis. In the Lithuanian sample, the ITQ had a good internal consistency with Cronbach's α of 0.86 (Dumarkaite et al., 2023).
The Resilience scale before intervention | Baseline
  Resilience before intervention is measured. The Resilience scale (RS-14, Wagnild, 2011) is a self-report measure comprising 14 items about resilience. All items are answered on a 7-point Likert scale that ranges from 1 (strongly disagree) to 7 (strongly agree). A higher score indicates more pronounced resilience. RS-14 will be used as a predictor in the analysis. The analysis of the psychometric properties of the RS-14 in the sample of Lithuanian adolescents demonstrated high reliability of the scale (Zelviene, 2020).
User satisfaction after intervention | Eight weeks after baseline
  The usability of the intervention is measured. Participants are asked to evaluate the usability of the intervention by indicating how useful (from 1 "not useful at all" to 5 "very useful"), satisfactory (from 1 "I did not like it at all" to 5 "I liked it a lot"), easy to use (from 1 "it was not easy at all" to 5 "it was very easy"), etc., the program is. Participants are also asked to report their subjective impression regarding the improvement of mental well-being (from 1 "worsened a lot" to 5 "improved a lot"), physical health (from 1 "worsened a lot" to 5 "improved a lot"), general understanding of oneself and one's well-being (from 1 "not at all" to 5 "definitely improved"), recommending the program to others (from 1 "not at all" to 5 "definitely would recommend"), etc.

CONTACTS AND LOCATIONS:
Overall Officials: Evaldas Kazlauskas, Ph.D., Principal Investigator — Vilnius University
Locations (1):
- Vilnius University, Vilnius, Vilnius County, Lithuania

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data can be shared upon a reasonable request.